

# STATISTICAL ANALYSIS PLAN

# FOR AC-055-303: SAP FOR CSR

SERAPHIN-OL: Study with an ERA in Pulmonary arterial Hypertension to Improve cliNical outcome (Open Label)

Long-term single-arm open-label extension study of the SERAPHIN study, to assess the safety and tolerability of macitentan/ACT-064992 in subjects with symptomatic pulmonary arterial hypertension

| Purpose of Analysis | Clinical Study Report |
|-----------------------|-----------------------|
| i dipose oi Aliaiysis | Chineal Study Report |

Investigational Drug JNJ-67896062/ACT-064992/Macitentan

Protocol Number AC-055-303

Document Number EDMS-RIM-297091

Document Status/Version Number Final

Date 21 December 2020

| PPD<br>PPD | , Statistician<br>, Expert Statistician |
|------------|-----------------------------------------|
| PPD | , Senior Clinical Leader |
| PPD | , Director Medical Safety Officer |
| PPD | , Director Medical Writing TA FL |
| PPD | , Senior Statistical Programmer |
| PPD | , Director, CTSL, Biometrics (SDS) |
| | PPD PPD PPD PPD |


The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.


# **TABLE OF CONTENTS**

| LIS | ST OF AI | ABBREVIATIONS AND ACRONYMS | 5 |
|---|---|---|---|
| 1 | INTRO | DDUCTION | 6 |
| 2 | STUDY | Y DESIGN AND FLOW | 6 |
| | 2.1<br>2.2 | Study design | |
| 3 | STUDY | Y OBJECTIVES | 12 |
| | 3.1<br>3.2 | Objectives for SERAPHIN DB | |
| 4 | | GES OR CLARIFICATIONS TO ANALYSES PLANNED Y PROTOCOL | |
| | 4.1<br>4.2<br>4.3 | Changes to the analyses planned in the study protocol<br>Changes in the conduct of the study / data collection<br>Clarifications concerning endpoint definitions and related | 13 |
| | - | statistical methods | |
| 5 | DEFINI | IITIONS OF VARIABLES | 13 |
| | 5.1<br>5.2<br>5.2 | Screening failures | 15 |
| | 5.2<br>5.2 | 2.2 Baseline disease characteristics | 16 |
| | | 2.4 Medical history | 16 |
| | | 5.2.5.1 Previous medications | 17 |
| | 5.3 | Study treatment exposure and compliance | 18 |
| | 5.3<br>5.3 | Compliance with study treatment | 19 |
| | 5.4<br>5.5 | Study discontinuation Efficacy variables | 19<br>19 |
| | 5.5 | 5.1 Long term survival | 19 |

# Confidential

| ZI December 2020, page 3/6 | 21 | December | 2020, | page | 3/6 |
|----------------------------|----|----------|-------|------|-----|
|----------------------------|----|----------|-------|------|-----|

| | 5.6 Safet | ty variables | 20 |
|---|---|---|---|
| | 5.6.1 | Adverse events | 20 |
| | 5.6.1 | .1 Treatment-emergent adverse events | ) |
| | 5.6.1 | .2 Frequency of treatment-emergent adverse events 20 | ) |
| | 5.6.1 | .3 Intensity of treatment-emergent adverse events | ) |
| | 5.6.1 | .4 Relationship of treatment-emergent adverse events 20 | ) |
| | 5.6.2 | Deaths | 21 |
| | 5.6.3 | Serious adverse events | 21 |
| | 5.6.4 | Adverse events leading to discontinuation of study treatment | 21 |
| | 5.6.5 | Other significant adverse events | 21 |
| | 5.6.6 | Vital signs and body weight | 21 |
| | 5.6.7 | Electrocardiogram | 21 |
| | 5.6.8 | Laboratory | 21 |
| | 5.6.8 | $\mathcal{C}_{\mathcal{I}}$ | |
| | 5.6.8 | $\sim$ | |
| | 5.6.8 | Incidence of abnormal hemoglobin values | 3 |
| 6 | DEFINITION | OF PROTOCOL DEVIATIONS IN AC-055-303 | 23 |
| _ | | | |
| 7 | ANALYSIS S | SETS | 24 |
| | 7.1 Defin | nitions of analysis sets | 24 |
| | 7.1.1 | Safety analysis set | |
| | 7.1.1 | | 4 |
| | 7.1.1 | | |
| | 7.2 Usag | ge of the analysis set | 24 |
| 8 | DEFINITION | OF SUBGROUPS | 25 |
| 9 | GENERAL S | TATISTICAL METHODOLOGY | 26 |
| | 9.1 Over | all testing strategy | 26 |
| | | eral rules for data presentations | |
| | | lay of patients disposition, protocol deviations and analysis set | |
| | | Subject disposition | |
| | 9.3.2 | Protocol deviations | |
| | 9.4 Anal | yses of patient characteristics | |
| | 9.4.1 | Demographics | |
| | 9.4.2 | Baseline disease characteristics | |
| | 9.4.3 | Other baseline characteristics | |
| | 9.4.4 | Medical history | |
| | 9.4.5 | Previous and concomitant medications | |
| | 9.5 Anal | ysis of study treatment exposure and compliance | |


| 21 December 2020, page 4/69 | 21 | Decem | ber | 2020, | page | 4/69 |
|-----------------------------|----|-------|-----|-------|------|------|
|-----------------------------|----|-------|-----|-------|------|------|

| | 9.5.1 | Exposure | | 28 |
|---|---|---|---|---|
| | 9.5.2 | Compliance with study treatment | | 28 |
| | 9.6 Analys | sis of the exploratory efficacy variable(s) | | 28 |
| | 9.6.1 | Hypothesis and statistical model | | 28 |
| | 9.7 Analys | sis of safety variables | | 29 |
| | 9.7.1 | Adverse events | | 29 |
| | 9.7.2 | Deaths, other serious adverse events | | 29 |
| | 9.7.2.1 | | 29 | |
| | 9.7.2.2 | | | |
| | 9.7.2.3 | | 30 | |
| | 9.7.2.4 | Adverse events leading to study treatment | | |
| | | discontinuations | | |
| | 9.7.2.5 | Other significant adverse events | 31 | |
| | 9.7.3 | Laboratory tests | | 31 |
| | 9.7.4 | Incidence of abnormal liver tests (including unscheduled | | |
| | | visits) | | |
| | 9.7.5 | Incidence of abnormal hemoglobin values | | |
| | 9.7.6 | Other laboratory parameters | | 33 |
| 10 | GENERAL DE | FINITIONS AND DERIVATIONS | | 33 |
| 11 | HANDLING O | F MISSING/INCOMPLETE DATE AND TIME FIELDS | | 36 |
| 12 | LIST OF SUM | MARY TABLES, LISTINGS AND FIGURES | | 40 |
| | 12.3.1 | Demographics and Patient Characteristics | | 40 |
| | 12.3.2 | Previous and concomitant therapies | | |
| | 12.4.1 | Exposure | | |
| | 12.5.1 | Adverse events | | 42 |
| | 12.5.2 | Deaths | | 43 |
| | 12.5.3 | Time to death | | 43 |
| | 12.5.4 | Serious adverse events | | 44 |
| | 12.5.5 | Adverse events leading to treatment discontinuation | | 44 |
| | 12.5.6 | Other significant adverse events | | |
| 13 | REFERENCES | | | 47 |
| 14 | APPENDICES. | | | 48 |


# LIST OF ABBREVIATIONS AND ACRONYMS

| AE | Adverse event |
|---------|----------------------------------------------|
| AESI | Adverse events of special interest |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| CRF | Case report form |
| CL | Confidence limit(s) |
| CSR | Clinical study report |
| DB | Double Blind |
| DOD | Date of death |
| eCRF | Electronic case report form |
| EOS | End-of-study |
| EOT | End-of-treatment |
| Hgb | Hemoglobin |
| KM | Kaplan-Meier |
| MedDRA | Medical Dictionary for Regulatory Activities |
| OL | Open label |
| PAH | Pulmonary arterial hypertension |
| PT | Preferred Term |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SAS | Statistical analysis system |
| SOC | System organ class |
| STRT302 | first dosing date in SERAPHIN DB |
| STRT303 | first dosing date in SERAPHIN OL |
| TEAE | Treatment-emergent Adverse Event |
| ULN | Upper limit of the normal range |
| WHO | World Health Organization |

## 1 INTRODUCTION

This Statistical Analysis Plan (SAP) details the final analysis conducted for the purpose of the production of the clinical study report (CSR) for the open-label (OL), extension study AC-055-303 (SERAPHIN OL) to the double-blind study AC-055-302 (SERAPHIN DB). This SAP also provides a description of the general considerations and assumptions, as well as the proposed list of tables, figures and listings for the pooled data of AC-055-302 (SERAPHIN DB) and AC-055-303 (SERAPHIN OL).

The pooling of AC-055-302 (SERAPHIN DB) and AC-055-303 (SERAPHIN OL) means that the data from the same patients randomized in SERAPHIN DB will be concatenated with their data from the OL extension study (SERAPHIN OL). The concatenation of data from the same patients is referred to as 'pooling' in this document.

The pooling will be done only for the survival and safety data of patients initially randomized to the Macitentan 10 mg dose in the SERAPHIN DB, up to the end of the study (if they did not participate in the SERAPHIN OL study) or end of SERAPHIN OL.

This SAP (unless explicitly specified) follows the derivations and conventions defined in the SERAPHIN DB SAP (AC-055-302 Analysis Plan, appendix 16.1.9 to AC-055-302 [SERAPHIN DB] CSR [D-12.425]).

### 2 STUDY DESIGN AND FLOW

### 2.1 Study design

A short summary of study design and its graphical presentation for AC-055-302 (SERAPHIN DB) and AC-055-303 (SERAPHIN OL) study are presented below.

**SERAPHIN DB** was a multicenter, randomized, double-blind, placebo-controlled, parallel group, event-driven Phase III study that compared oral once daily treatment with 3 mg and 10 mg doses of Macitentan versus placebo in patients with symptomatic pulmonary arterial hypertension (PAH).

Patients aged 12 years or over were eligible to be enrolled if diagnosed with World Health Organization (WHO) FC II—IV idiopathic PAH, familial PAH, PAH associated with connective tissue disease, PAH associated with simple congenital systemic-to-pulmonary shunts at least 1-year post-surgical repair, HIV infection, or drugs and toxins.

A total of 742 patients were randomized in a 1:1:1 ratio to Macitentan 3 mg (n = 250), Macitentan 10 mg (n = 242), and placebo (n = 250) in SERAPHIN DB.

The study took place from 25 May 2008 (first subject/first visit) until 15 March 2012 (last subject/last visit).


The Macitentan 10 mg treatment effect (active vs. placebo) was highly statistically significant and clinically relevant, with a hazard ratio for the composite endpoint (Death; Atrial septostomy; Lung transplantation; Initiation of intravenous (i.v.) or subcutaneous prostanoids; Other worsening of PAH) of 0.547 (97.5% confidence limits [CLs] 0.392, 0.762, logrank p < 0.0001). More details are available in the Clinical Study Report (D-12.425). The Macitentan 10 mg daily dose was approved by European Medicines Agency, Food and Drug Administration, and most other regulatory authorities around the world.

Patients who prematurely discontinued study treatment (DB) due to clinical worsening of PAH and obtained written approval from Actelion, and patients who completed the study as scheduled, could enter SERAPHIN OL. For patients who had opted not to participate or who were not eligible to participate in SERAPHIN OL a 28-day safety follow-up after end of treatment (EOT) was performed.

**SERAPHIN OL** is an open-label, non-comparative, multicenter, extension study to assess long-term safety and tolerability of Macitentan in patients with symptomatic PAH, who either completed the DB treatment period of SERAPHIN or had clinical worsening of PAH in SERAPHIN. The OL study enrolled 550 patients (first patient enrolled on 17 October 2008), all of whom received Macitentan 10 mg, irrespective of DB treatment allocation.

The study treatment period for each patient lasts from his/her enrollment date until the end of the trial defined as the earliest of:

- (i) approval of Macitentan in this indication is obtained in the patient's country,
- (ii) the sponsor decides to stop study AC-055-303 (SERAPHIN OL),
- (iii) the subject's, investigator's, or sponsor's decision to discontinue study drug.


# Figure 1 AC-055-302 (SERAPHIN DB) and AC-055-303 (SERAPHIN OL) study design

Figure 1 Study design



Table 1 All patients treated in SERAPHIN DB (AC-055-302) and/or SERAPHIN OL (AC-055-303)

| Study number (Acronym) | randor<br>Macitent<br>AC-0<br>(SERAF | of patients<br>mized to<br>an 3 mg in<br>55-302<br>PHIN DB) | randon<br>Maciten<br>in AC-<br>(SERAF | of patients<br>mized to<br>tan 10 mg<br>055-302<br>PHIN DB)<br>= 242 | Number of patients randomized to placebo in in AC-055-302 (SERAPHIN DB) N = 250 | | Epatients in<br>SERAPHIN<br>N= 550 | |
|---|---|---|---|---|---|---|---|---|
| AC-055-302<br>(SERAPHIN<br>DB)<br>treatment /<br>AC-055-303<br>(SERAPHIN<br>OL)<br>treatment | 3 mg /<br>none:<br>N = 65 | 3 mg /<br>10 mg:<br>N = 185 | 10 mg /<br>none:<br>N = 60 | 10 mg /<br>10 mg:<br>N = 182 | Placebo /<br>10 mg:<br>N = 183 | Placebo /<br>10 mg:<br>N = 183 | 3 mg /<br>10 mg:<br>N = 185 | 10 mg /<br>10 mg:<br>N =<br>182 |

DB = double-blind, OL = open-label.

Patients who did not enter the open-label study are shown in the columns '3 mg / none' and '10 mg / none'. Those who received Macitentan in both the double-blind and open-label periods are shown in the '3 mg / 10 mg' and '10 mg' and '10 mg' columns. Finally, those who received placebo in the double-blind study and entered the extension study are shown in the 'Placebo / 10 mg' column.

Analyses will be provided for the following cohorts (see below and Table 2):

- Macitentan 10 mg OL (550 patients): This cohort comprises all patients enrolled into SERAPHIN OL who took at least one dose of Macitentan 10 mg as an OL treatment (regardless of randomized treatment in SERAPHIN DB). As this group is heterogenous (initially the patients were randomized to different treatment regimens) it will be further analyzed by randomization groups.
  - o Placebo DB/Macitentan 10 mg OL (183 patients)
  - o Macitentan 3 mg DB/Macitentan 10 mg OL (185 patients)
  - o Macitentan 10 mg DB/Macitentan 10 mg OL (182 patients)
- Macitentan 10 mg DB/OL (242 patients): This cohort comprises all patients randomized to Macitentan 10 mg in SERAPHIN DB. For this group of patients, data from SERAPHIN DB and SERAPHIN OL will be pooled within patient.

**Table 2** Template for summary tables

| | Macitentan 10 mg (OL) | | | |
|---|---|---|---|---|
| Macitentan 10 mg<br>(DB/OL) | Placebo /<br>10 mg:<br>(N = 183) | 3 mg /<br>10 mg:<br>(N = 185) | 10 mg /<br>10 mg:<br>(N = 182) | Total<br>(N=550) |
| (N=242) | | | | |


# 2.2 Study Visit and Assessment Schedule

# Table 3 Visit and Assessment Schedule for Seraphin DB

Table 1 Visit and assessment schedule

| 1 able 1 | visit and as | ssessment schedu | пе | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| PERIODS | SCREENING | | TREATMENT PERIOD FOLLOW-UP PER | | | | | | UP PERIOD | |
| VISITS | 1 | 2 | 3 | 4 | 5 | 6, 7 etc. | EVENT | End-of-Treatment | End-of-Study9 | Follow-up |
| | Screening | Randomization | | | | | | (EOT) | (EOS) | - |
| TIME POINTS | Day -28 to -1 | Day 1 | Month 3 | Month 6 | Month 12 | Every 6 | | Study drug | Target number | 28 days after |
| | | | ± 2 weeks | ±2 weeks | ±2 weeks | months | | discontinuation | of events | study drug |
| ASSESSMENTS | | | | | | <u>+</u> 2 weeks | | | achieved | discontinuation |
| Informed consent | X | | | | | | | | | |
| Medical history | X | | | | | | | | | |
| Concomitant medications | X | X | X | X | X | X | X | X | | |
| Vital Signs, body weight | X | X | X | X | X | X | X | X | | |
| 12-lead ECG | X | | | X | | | X <sup>8</sup> | X | | |
| Complete laboratory tests <sup>1</sup> | X | | X | X | X | X | $X^8$ | X | | |
| LFTs and PK sampling (serum) <sup>10</sup> | | | | M | lonthly (+/- 1 v | veek) monito | ring up to a | t least 28 days after En | d-of-Treatment | |
| Pregnancy Test <sup>2</sup> | X | $X^3$ | | , | Monthly (+/ | - 1 week) and | up to at lea | st 28 days after End-o | f-Treatment | |
| NT-pro-BNP | | X | | X | | | | | | |
| Right heart catheterization | | X <sup>4</sup> | | $X^5$ | | | | | | |
| Modified WHO class | X | X | X | X | X | X | X | X | | |
| 6MWT | X | X | X | X | X | X | X | X | | |
| Borg dyspnea index | X | X | X | X | X | X | X | X | | |
| PK sampling (plasma) | | | | $X^5$ | | | $X^8$ | X | | |
| QoL questionnaire (SF 36) | | X | | X | X | | X <sup>8</sup> | X | | |
| Study drug dispensing | | X | | X | X | X | | | | |
| Adverse events <sup>6</sup> | | X | X | X | X | X | X | X | | X |
| Serious adverse events <sup>6</sup> | $X^7$ | X | X | X | X | X | X | X | | X |
| Vital status | | | | | | | | | X | |

<sup>&</sup>lt;sup>4</sup> Includes hematology and chemistry, <sup>3</sup> Women of childbearing potential only, <sup>3</sup> Urine-dipstick pregnancy test if last negative serum pregnancy test older than 2 weeks; <sup>4</sup> Only to be performed if not done within 12 months (3 months for patients participating in the PK/PD sub-study, <sup>6</sup> AE and SAE reporting and follow-up: all AEs/SAEs from study drug initiation up to 28 days after study drug discontinuation, follow-up of ongoing AEs/SAEs only thereafter, <sup>7</sup> SAE reporting: during screening period, SAEs related to study-mandated procedures only, <sup>8</sup> Only if event leads to study drug discontinuation; <sup>9</sup> EOS Visit will coincide with EOT Visit if patient completes the study as scheduled; <sup>10</sup> PK in serum is only to be analyzed at EOS if liver aminotransferases is above 3 times ULN.


# Table 4 Visit and Assessment Schedule for Seraphin OL

| PERIODS | | TREATMENT PERIOD | | |
|---|---|---|---|---|
| VISITS | Enrolmnent (Visit 1) | Visit 2,3, etc. | End-of-Treatment (EOT) | End-of-Study (EOS) |
| TIMEPOINTS | Day 1 <sup>1</sup> | Month 6,<br>and every 6 months<br>thereafter | Up to 28 days after study drug discontinuation | |
| ASSESSMENTS | | $\pm 2$ weeks | | |
| Informed Consent | X | | | |
| Concomitant medication | X | X | X | X |
| Vital signs, Body weight Physical examination | Performed at ea | each visit; Data will only be kept in patient's file | | |
| Complete Laboratory Tests | X | X | X | |
| LFTs | X | Recommended monthly (+/-1 week) | | |
| LITS | Λ | up to at least 28 days after End-of-Treatment | | |
| Serum Pregnancy Test <sup>2</sup> (if applicable) | X | X | | |
| Urine Pregnancy Test <sup>2,5</sup> | | | Required monthly (+/-1 wee | k) |
| (if applicable) | | up t | o at least 28 days after End-of-T | reatment |
| Phone call for pregnancy test | | | Required monthly (+/-1 wee | k) |
| reminder and contraception | | up to at least 28 days after End-of-Treatment | | |
| Study Drug Dispensing <sup>4</sup> | X | X | | |
| Adverse Events <sup>3</sup> | X | X | X | X |
| Serious Adverse Events | X | X | X | X |

<sup>1</sup>The tests are not to be repeated if measured during the End-of-Treatment visit of study AC-055-302/SERAPHIN that has been performed within 4 weeks of this visit. <sup>2</sup>Women of childbearing potential only; <sup>3</sup>AE reporting and follow-up: all AEs up to 28 days after study drug discontinuation. <sup>4</sup>Study drug may be dispensed on a monthly basis at each LFT visit. <sup>5</sup>Urine pregnancy test is required if no serum pregnancy test is performed. AE = adverse event; LFT = liver function test.


### 3 STUDY OBJECTIVES

# 3.1 Objectives for SERAPHIN DB

# **Primary objective**

The primary objective of this study was to demonstrate that either dose (3 mg or 10 mg) of Macitentan reduces the risk of morbidity and mortality in patients with symptomatic PAH.

## Secondary objectives

- To demonstrate that either dose (3 mg or 10 mg) of Macitentan improves exercise capacity, WHO FC, and reduces the risk of death due to PAH or hospitalization for PAH up to end-of-treatment (EOT) in patients with symptomatic PAH.
- To demonstrate that either dose (3 mg or 10 mg) of Macitentan reduces the risk of death of all causes up to EOT and up to end-of-study (EOS).
- To evaluate the safety and tolerability of Macitentan in patients with symptomatic PAH

# 3.2 Objectives for SERAPHIN OL

To assess long-term safety and tolerability of Macitentan in patients with symptomatic PAH.

# 4 CHANGES OR CLARIFICATIONS TO ANALYSES PLANNED IN THE STUDY PROTOCOL

# 4.1 Changes to the analyses planned in the study protocol

This SAP was prepared based on the Protocol AC-055-303 OL version 7 (17 July 2020).

For the two cohorts described in section 2.1, the Safety Set is defined as:

Macitentan 10 mg DB/OL - all patients who received at least one 10 mg dose of Macitentan in DB/OL and with at least one post-baseline assessment.

Macitentan 10 mg OL (550) - all patients who were enrolled and received Macitentan in SERAPHIN OL study.

For details for safety set see Section 7.1.1.

Laboratory data will not be normalized but presented as collected.

Mean daily dose is not analyzed as most patients treated with Macitentan received 10 mg (610/675 = 90%) patients, where 675 is number of patients who received Macitentan either in DB or OL period).

Statistical Analysis Plan EDMS-RIM-297091

In the protocol no primary efficacy endpoint was defined for this OL extension study. However, long-term survival can be evaluated for those patients that entered the study, as well as for the pooled DB/OL cohort as defined above.

# 4.2 Changes in the conduct of the study / data collection

---

# 4.3 Clarifications concerning endpoint definitions and related variables or statistical methods

For the Macitentan 10 mg DB/OL cohort, time to death will be calculated using start of the Macitentan 10 mg treatment at the beginning of dosing in DB period. Full details for time to event analysis are given in section 5.5.1.

In this SAP the per-protocol dataset is not defined. Protocol deviations will be reported as per section 6.

Adverse events of special interest were not pre-specified in the protocol. They are defined in section 5.6.5.

Table 2 defines the cohorts to be presented for the summaries.

## 5 DEFINITIONS OF VARIABLES

The following dates will be used to define the treatment durations, survival, censoring and safety reporting periods: For imputation of partial/missing date, refer to section 11.

- Start date of Macitentan in SERAPHIN DB (STRT302): date of first administration of Macitentan in patients randomized to Macitentan 10 mg in SERAPHIN DB collected in the study drug log.
- Enrollment date into SERAPHIN OL (STRT303): date of enrollment into SERAPHIN OL as reported in the Interactive Voice Response System (IVRS) system.
- Date of death (DOD): actual date of death of a patient as reported in the SERAPHIN DB or SERAPHIN OL Case Report Forms (CRFs) prior to the SERAPHIN OL study closure.
- CENS: Censoring flag. Categorical: 0 (not censored) or 1 (censored).


• **SERAPHIN DB End Of Study (EOS302)**: This is the end of study (EOS) visit date of a patient from the SERAPHIN DB study.

Note that for all patients who did not withdraw prematurely from SERAPHIN DB, the **EOS302** occurred shortly after the administrative end of SERAPHIN DB announced by Actelion on 30 January 2012.

• SERAPHIN OL EOS (EOS303): study completion date.

Note that the end of the study in SERAPHIN OL is on a patient-by-patient basis, until the earliest between:

- o Death
- The latest date between: Date of visit/ Contact or Date of discontinuation/ Last contact on the EOS/Permanent Discontinuation CRF page.

The EOS occurs when the approval of Macitentan is obtained in the patient's country or when the patient, investigator, or sponsor decides to discontinue study drug.

EOS302 and EOS303 (individual patient's end of study) will be referred in this SAP as end of study (EOS). The overall end of study up to the database lock will be referred as study closure.

- End of Treatment in SERAPHIN DB (EOT302): end of double-blind treatment in SERAPHIN DB, i.e., the last treatment date reported in the SERAPHIN DB study drug log.
- End of Treatment in SERAPHIN OL (EOT303): EOT in SERAPHIN OL, i.e., the last treatment end date reported in the study drug log.
- **SERAPHIN OL last contact date (LAST303)** No ongoing patients are expected anymore, therefore LAST303=EOS303
- **SERAPHIN DB last contact date (LAST302)** No ongoing patients are expected anymore, therefore LAST302=EOS302
- Last contact date (LCTC) for SERAPHIN OL and DB: This is the latest date between LAST303 and EOS302. For patients who did not enter SERAPHIN OL, the date will be EOS302.
- EOT in SERAPHIN OL and DB:
  - o For patients in the OL cohort this is EOT303.
  - o For patients in the DB/OL cohort:
    - If the patient entered SERAPHIN OL then this is EOT303.


- If the patient did not enter SERAPHIN OL then this is EOT302.
- **Time to death (TTD)** is estimated by the Kaplan-Meier (KM) product limit method and summarized for each cohort, except Macitentan total (SAP for sNDA Section 6.1).

For example, for cohort Macitentan 10 mg DB/OL, time to death was defined as the time of start of Macitentan 10 mg treatment in SERAPHIN DB up to the date of death (any cause) in either the DB or OL period. Patients who did not die prior to the study closure were censored at their last date of contact.

For patients in the Macitentan 10 mg DB/OL cohort **who died prior to study closure**, time to death is derived:

TTD=DOD - STRT302 and CENS=0 and,

For patients in the Macitentan 10 mg DB/OL cohort who did not die prior study closure and therefore censored:

TTD=LCTC - STRT302 and CENS=1 Where LCTC=max(EOS302, EOS303).

Imputation rules for missing or incomplete dates are listed in section 11.

# 5.1 Screening failures

Not Applicable for this SAP.

## 5.2 Patients characteristics

Baseline information for the patients in the Macitentan 10 mg OL cohort is defined as the latest available information prior to the first dosing date in the OL study.

Baseline information for patients in the Macitentan 10 mg DB/OL cohort is defined as the latest available information prior to the first dosing date in SERAPHIN DB (STRT302).

For patients in the Macitentan 10 mg DB/OL cohort, completion/discontinuation of study drug and the associated reasons will be counted either in SERAPHIN DB if the patients did not enter SERAPHIN OL (10 mg / none), or in SERAPHIN OL if the patients entered SERAPHIN OL (10 mg / 10 mg).

For patients in Macitentan 10 mg OL cohort, completion/discontinuation of study drug and associated reasons will be counted in SERAPHIN OL.

The study drug discontinuation rate will be adjusted on person-year of study duration for each cohort and each drug dose sequence.


# 5.2.1 Demographics

Demographics will include: age (years), age subgroups (Adolescents [< 18 years], from 18 to 64 years, from 65 to 84 years, and over 84 years), gender (Male, Female), race (White [including Hispanic], Asian, Other), height (cm), weight (kg) and body mass index (BMI; kg/m²), geographical location (North America including Canada; Western Europe including South Africa and Israel; Eastern Europe including Turkey; Asia including Australia; Latin America).

Age (years) = (STRT303 - birth date + 1)/365.25 will be reported as number of completed years.

For the Macitentan 10 mg DB/OL, age is the age at the first dose in DB.

For the Macitentan 10 mg OL, age is the age at entry into OL.

For imputation of partial birth date, refer to section 11.

#### **5.2.2** Baseline disease characteristics

Baseline disease characteristics will include PAH etiology at baseline (idiopathic, familial, associated with HIV infection, associated with drug use or toxin exposure, associated with collagen vascular disease, associated with repaired congenital shunts) and WHO FC at baseline.

## 5.2.3 Other baseline characteristics

Other baseline characteristics will include categorized Estimated Creatinine Clearance:

- no renal impairment (creatinine clearance  $\geq 90 \text{ mL/min}$ ),
- mild renal impairment (creatinine clearance  $\geq 60$  and < 90 mL/min)
- moderate-severe renal impairment (creatinine clearance < 60 mL/min).

### **5.2.4** Medical history

Medical History is not summarized for this analysis as it was previously reported for the CSR of AC-055-302 (SERAPHIN DB).

#### 5.2.5 Previous and concomitant medications

Previous and concomitant medications for SERAPHIN DB and SERAPHIN OL are coded using WHO Drug Dictionary version March 2019.

In SERAPHIN OL, collection in the CRF of previous and concomitant medications was introduced with Global Protocol Amendment 4 (27 August 2013). Medications taken prior to implementation of this protocol amendment were then collected retrospectively. Medications which were 'ongoing at EOT' in the SERAPHIN DB are reconciled with medications 'ongoing at the start of AC-055-303' (SERAPHIN OL). Since the SERAPHIN DB was closed prior to the retrospective data collection, any discrepancies identified in


Statistical Analysis Plan EDMS-RIM-297091

this database cannot be corrected. These discrepancies are reported in a Data Management tracker by the Global Data Manager, and will be reported in a separate listing.

Patients who took the same medication more than once (as qualified by the same preferred term (PT) will be counted only once. In case the reported medication was assigned to several PTs, patients are counted for each individual PT.

#### 5.2.5.1 Previous medications

A previous medication is any treatment for which the end date of treatment is prior to the start of the AC-055-303 (SERAPHIN OL) study (i.e., prior to signing the informed consent form). These are not included in the analysis as these are part of the AC-055-302 (SERAPHIN DB) CSR; these data were reported as previous or concomitant therapies.

#### 5.2.5.2 Concomitant medications

Concomitant medications are all treatments that are ongoing or initiated after start of study (i.e., from the time of the patient signing the informed consent form) or initiated up to 28 days after the end of study treatment.

Concomitant medication at baseline is defined as any medication that is taken at the start of study drug (STRT303 for Macitentan 10 mg OL, STRT302 for Macitentan 10 mg DB/OL). This includes any medication with the tick box "ongoing at Baseline" checked, or with a start date before or on the day of study drug start (STRT303 for Macitentan 10 mg OL, STRT302 for Macitentan 10 mg DB/OL) and the end date not before study drug start (STRT303 for Macitentan 10 mg OL, STRT302 for Macitentan 10 mg DB/OL). Start and end dates that are incomplete will be handled according to the rules for partial and missing concomitant medication dates in section 11 **Appendix A**.

Note: the concomitant medications at baseline for patients in the Macitentan 10 mg DB/OL cohort will be derived using only the AC-055-302 (SERAPHIN DB) database. For patients in the Macitentan 10 mg OL cohort, both AC-055-302 (SERAPHIN DB) and AC-055-303 (SERAPHIN OL) databases will be used for the derivation of concomitant medications at baseline.

# PAH therapies

PAH therapy includes phosphodiesterase-type 5 (PDE-5) inhibitors, prostanoids, and soluble guanylate cyclase stimulators, and comprises the following PT:

- PDE-5 inhibitors, including:
  - o Sildenafil
  - o Tadalafil
  - o Vardenafil
- Drugs acting via prostacyclin pathway / prostanoids, including
  - Iloprost
  - Beraprost


- o Treprostinil
- o Epoprostenol
- o Selexipag
- Soluable guanylate cyclase stimulators, including:
  - o Riociguat

In the medication selection for PAH therapy, any medication coded PT that contains one of the PT included in the definition above is used (e.g. "sildenafil citrate" is a PAH specific medication that belongs to the PDE-5 inhibitor category.)

Concomitant medications during the study include all concomitant medications at baseline plus the medication reported as 'ongoing at end of treatment/study' or with the start date on or after the start date of study drug treatment:

- STRT302 for Macitentan 10 mg [DB/OL],
- STRT303 for Macitentan 10 mg [OL]

and on or before the EOT+28 days.

The following summaries will be presented for each cohort:

• A summary of concomitant PAH therapy at baseline (for baseline DB and separately baseline OL) including the number and percentages of patients taking at least one PAH therapy (i.e., at least one PDE-5 inhibitor, at least one prostanoid).

Note: patients may receive more than one treatment and may be included in more than one treatment class.

- A summary of concomitant medication use at baseline for all medications taken by at least 5.0% patients in any cohort, by PT
- A summary of concomitant medication use during the study for all medications taken by at least 5.0% in any cohort, by PT.

A listing of concomitant medications will be provided.

# 5.3 Study treatment exposure and compliance

## 5.3.1 Exposure

The duration of treatment (exposure) is defined as the time from start of dosing of Macitentan 10 mg (for the Macitentan 10 mg DB/OL mg cohort it is from STRT302, for the Macitentan 10 mg OL cohort it is from STRT303) until EOT inclusive, regardless of treatment interruptions.


Duration of treatment exposure will be calculated by cohort as follows:

Duration (days) = EOT303 - STRT303 +1, for patients in the Macitentan 10 mg OL,

or

Duration (days) = max(EOT302, EOT303) - STRT302 +1, for patients in the Macitentan 10 mg DB/OL.

Duration (months) = Duration (days)  $\sqrt{30.4375}$ 

# **5.3.2** Compliance with study treatment

Not Applicable

## 5.3.3 Study treatment discontinuation

Study treatment discontinuations include all patients, i.e., those who prematurely discontinued and those who completed treatment as per protocol, from eCRF study Drug log.

Reasons for study treatment discontinuation are retrieved from the study drug log CRF pages in SERAPHIN DB or OL as appropriate and are coded using Actelion Study Drug Log dictionary.

## 5.4 Study discontinuation

Study completion/discontinuation is collected in the eCRF study completion page.

## 5.5 Efficacy variables

### 5.5.1 Long term survival

Time to death (TTD; in months) in the two cohorts is defined as follows:

For the Macitentan 10 mg OL cohort:

TTD (in days) and censoring flag (CENS) will be derived using the dates defined as:

- TTD = DOD STRT303 and CENS = 0 for patients who died,
- TTD = LCTC STRT303 and CENS = 1 for patients who did not die.

For the Macitentan 10 mg DB/OL cohort:

- TTD = DOD STRT302 and CENS = 0 for patients who died,
- TTD = LCTC STRT302 and CENS = 1 for patients who did not die.


For both cohorts

TTD (in months) = TTD (in days) / 30.4375.

Patients censored will be those who did not die prior to study closure.

## 5.6 Safety variables

AEs are coded using MedDRA v.21.0. For imputation of AE onset/resolution date, refer to Section 11.

## 5.6.1 Adverse events

## 5.6.1.1 Treatment-emergent adverse events

Treatment-emergent adverse events (TEAEs) are defined as AEs occurring during Macitentan OL treatment period (defined in section 10) for the Macitentan 10 mg OL cohort and during the Macitentan DB/OL treatment period (defined in section 10) for the Macitentan 10 mg DB/OL cohort (see section 10), with onset date ≥ start date (STRT302 for Macitentan 10 mg [DB/OL], STRT303 for Macitentan 10 mg [OL]), and up to 28 days (inclusive) after EOT. Note: if AEs are recorded before STRT303, these AEs will not be included for Macitentan 10 mg (OL) cohort.

# 5.6.1.2 Frequency of treatment-emergent adverse events

Treatment-emergent AEs reported more than once by a patients will be counted only once in the frequency tables.

In the event that the reported TEAE is assigned to several PT, patients will be counted for each individual PT.

# 5.6.1.3 Intensity of treatment-emergent adverse events

The categories of intensity are defined as follows:

- Mild
- Moderate
- Severe

For TEAEs reported more than once for a patient within a specified analysis time period but with different intensities, the worst intensity is considered (i.e. severe). If intensity is missing, the event will be considered to be severe.

## 5.6.1.4 Relationship of treatment-emergent adverse events

Relationship to study treatment is defined as 'related' or 'not related' in the opinion of the investigator. For TEAEs reported more than once for a patients within the same time period, the worst relationship will be used (i.e. 'related'). Adverse events with missing relationships will be considered in any analysis to be 'related'.


Statistical Analysis Plan EDMS-RIM-297091

#### **5.6.2** Deaths

Cause of death is derived as collected on the disposition CRF page. There can be more causes of death recorded per patient. All reported causes of death will be used.

#### **5.6.3** Serious adverse events

SAEs refer to AEs qualified as "serious" by the investigator on the CRF AE page(s). If seriousness information is missing, then AEs will be summarized as 'Serious AEs' (the worst-case scenario).

# 5.6.4 Adverse events leading to discontinuation of study treatment

Adverse events leading to discontinuation of study treatment are those with an action taken with study drug of "permanently discontinued" recorded on the CRF AE page.

# 5.6.5 Other significant adverse events

AEs of special interest are defined using selection of PTs (Actelion Internal MedDRA Query). The selection is defined from medical review of terms in the MedDRA v. 21.0 dictionary and where applicable, Standardized MedDRA Queries (SMQs) were used (see SMQ Introductory Guide Version 19.1: September 2016 – MMSO-DI-6226-19.1.0). The full definition is included in Appendix C.

The following groups of AEs of special interest will be summarized:

- o liver abnormalities,
- o edema.
- o anemia/ hemoglobin decrease,
- o hypotension.

### 5.6.6 Vital signs and body weight

Not Applicable

### 5.6.7 Electrocardiogram

Not Applicable

### 5.6.8 Laboratory

All available laboratory data collected at local and central laboratory will be used for deriving laboratory abnormalities.

Baseline laboratory values are defined as the latest values recorded before or on the date of first dose of Macitentan for DB/OL and for OL before or on the date of first dose of Macitentan in OL. Treatment-emergent values are defined as post-baseline values occurring within EOT+28 days and will be considered in the tables.


# 5.6.8.1 Hematology and blood chemistry

Hematology and blood chemistry tests include hemoglobin, hematocrit, platelet, leukocyte, and erythrocyte counts, liver aminotransferases (AST/ALT), alkaline phosphatase, total and direct bilirubin, creatinine, urea, glucose, sodium, potassium and albumin.

Marked laboratory abnormalities are defined according to Actelion internal guidelines for individual parameters (see Table ).

**Table 5** Laboratory Abnormalities

| Parameter | LL marked | LLL marked | HH marked | HHH marked |
|---|---|---|---|---|
| Hemoglobin | < 100 g/L | < 80 g/L | post-baseline > (baseline + 20 g/L) | post-baseline > (baseline + 40 g/L) |
| Hematocrit | < 0.28 L/L for females | < 0.20 L/L | > 0.55 L/L for females | > 0.65 L/L |
| | < 0.32 L/L for males | | > 0.60 L/L for males | |
| Platelets | $< 75 \times 10^{9}/L$ | $< 50 \times 10^{9}/L$ | $> 600 \times 10^9 / L$ | $> 999 \times 10^9/L$ |
| Leukocytes | $< 3.0 \times 10^{9}/L$ | $< 2.0 \times 10^9/L$ | $> 20.0 \times 10^9/L$ | $> 100.0 \times 10^9/L$ |
| Lymphocytes | $< 0.8 \times 10^{9}/L$ | $< 0.5 \times 10^9 / L$ | $> 4.0 \times 10^9 / L$ | $> 20 \times 10^{9}/L$ |
| ALT | NA | NA | > 3 × ULN | > 5 × ULN* |
| AST | NA | NA | > 3 × ULN | > 5 × ULN* |
| Alkaline<br>phosphatase | NA | NA | > 2.5 × ULN | > 5 × ULN |
| Total Bilirubin | NA | NA | > 2 × ULN | > 5 × ULN |
| Creatinine | NA | NA | > 1.5 × ULN | $> 3 \times ULN$ |
| Glucose | < 3.0 mmol/L | < 2.2 mmol/L | > 8.9 mmol/L | > 13.9 mmol/L |
| Calcium | < 2.0 mmol/L | < 1.75 mmol/L | > 2.9 mmol/L | > 3.1 mmol/L |
| Sodium | NA | < 130 mmol/L | > 150 mmol/L | > 155 mmol/L |
| Potassium | < 3.2 mmol/L | < 3.0 mmol/L | > 5.5 mmol/L | > 6.0 mmol/L |
| Albumin | < 30 g/L | < 20 g/L | NA | NA |

<sup>\*</sup> Also HHHH as > 8 × ULN

ALT = alanine aminotransferase; AST = aspartate aminotransferase; NA = not applicable/available; ULN = upper limit of normal.


# 5.6.8.2 Abnormal liver tests (including unscheduled visits)

Hepatic abnormality criteria are specified below:

- (ALT  $\geq$  3 × upper limit of normal [ULN]) **OR** (AST  $\geq$  3 × ULN)
- (ALT  $\geq$  5 × ULN) **OR** (AST  $\geq$  5 × ULN)
- (ALT  $\geq$  8 × ULN) **OR** (AST  $\geq$  8 × ULN)
- Total Bilirubin > 2 × ULN
- $\{(ALT \ge 3 \times ULN) \ \mathbf{OR} \ (AST \ge 3 \times ULN)\} \ \mathbf{AND} \ (Total \ Bilirubin \ge 2 \times ULN \ at \ any \ time)$

For each patient, the worst treatment-emergent abnormal value (i.e., the highest ALT, AST or Total Bilirubin values) will be considered and assigned to the appropriate category (may be more than one category per patient).

## 5.6.8.3 Incidence of abnormal hemoglobin values

Hemoglobin (Hgb) abnormalities are specified as:

- $Hgb \le 80 \text{ g/L}$
- $Hgb \le 100 \text{ g/L}$
- Hgb decrease from baseline  $\geq 20 \text{ g/L}$
- Hgb decrease from baseline  $\geq 50 \text{ g/L}$

For each patient, the worst treatment-emergent abnormal value (i.e., the lowest Hgb value) will be considered and assigned to the appropriate category (may be more than one category per patient).

Hgb abnormalities for increase from baseline are specified as:

- Post-baseline Hgb > (baseline + 20 g/L)
- Post-baseline Hgb > (baseline + 40 g/L)

For each patient, the worst treatment-emergent abnormal value (i.e., the highest Hgb value) will be considered and assigned to the appropriate category (may be more than one category per patient).

### 6 DEFINITION OF PROTOCOL DEVIATIONS IN AC-055-303

Protocol deviations will be reported as per Appendix E for the Macitentan 10 mg OL cohort.

### 7 ANALYSIS SETS

# 7.1 Definitions of analysis sets

## 7.1.1 Safety analysis set

The safety analysis set (SAF) will include all patients who received at least one dose of Macitentan 10 mg. All summaries described in this SAP will be presented on the SAF. Safety population will consist of the 2 cohorts described below.

# 7.1.1.1 Macitentan 10 mg OL cohort

This cohort includes 550 patients enrolled to the AC -055-303/SERAPHIN OL (regardless of the randomized treatment in SERAPHIN DB). As this group is heterogenous (initially the patients were randomized to different treatment regimens), so in addition to Overall, it will be further analyzed by randomization groups:

- o Placebo DB/Macitentan 10 mg OL (183 patients)
- o Macitentan 3 mg DB/Macitentan 10 mg OL (185 patients)
- o Macitentan 10 mg DB/Macitentan 10 mg OL (182 patients)

# 7.1.1.2 Macitentan 10 mg DB/OL cohort

This cohort includes 242 patients initially randomized to Macitentan 10 mg SERAPHIN DB. For this group of patients, information collected during SERAPHIN DB and SERAPHIN OL will be pooled within patient, meaning that the data from the same patients randomized in SERAPHIN DB will be concatenated with their data from the OL extension study (SERAPHIN OL).

# 7.2 Usage of the analysis set

**Table 6 Summaries by Analyses Cohorts.** 

| | | Macitentan 10 mg OL | | | |
|---|---|---|---|---|---|
| Summaries and analyses | Macitentan<br>10 mg<br>DB/OL<br>(N = 242) | Placebo<br>DB/<br>Macitentan<br>10 mg OL<br>(N = 183) | Macitentan<br>3 mg DB/<br>Macitentan<br>10 mg OL<br>(N =185) | Macitentan<br>10 mg DB/<br>Macitentan<br>10 mg OL<br>(N = 182) | Macitentan<br>10 mg OL<br>Total<br>(N = 550) |
| Disposition of patients | Yes | Yes | Yes | Yes | Yes |
| Demographics and patient characteristics | Yes | Yes | Yes | Yes | Yes |
| Medical history of patients | No | No | No | No | No |


| | | Macitentan 10 mg OL | | | |
|---|---|---|---|---|---|
| Summaries and analyses | Macitentan<br>10 mg<br>DB/OL<br>(N = 242) | Placebo<br>DB/<br>Macitentan<br>10 mg OL<br>(N = 183) | Macitentan<br>3 mg DB/<br>Macitentan<br>10 mg OL<br>(N =185) | Macitentan<br>10 mg DB/<br>Macitentan<br>10 mg OL<br>(N = 182) | Macitentan<br>10 mg OL<br>Total<br>(N = 550) |
| Concomitant<br>Medication | Yes | Yes | Yes | Yes | Yes |
| Duration of<br>Treatment exposure | Yes | Yes | Yes | Yes | Yes |
| Adverse events (AEs) | Yes | Yes | Yes | Yes | Yes |
| Serious Adverse<br>Events (SAEs) | Yes | Yes | Yes | Yes | Yes |
| AEs of special<br>interest* (as per<br>Actelion Internal<br>MedDRA Queries<br>[AIMQ]) | Yes | Yes | Yes | Yes | Yes |
| Deaths | Yes | Yes | Yes | Yes | Yes |
| AEs leading to permanent discontinuation of study treatment | Yes | Yes | Yes | Yes | Yes |
| Incidence of AEs over time | Yes | Yes | Yes | Yes | Yes |
| Incidence of abnormal liver test | Yes | Yes | Yes | Yes | Yes |
| Incidence of abnormal hemoglobin test | Yes | Yes | Yes | Yes | Yes |
| Time to Death<br>(Survival Analysis<br>using KM<br>approach) | Yes | Yes | Yes | Yes | Yes |

AE = adverse event, AIMQ = Actelion Internal MedDRA Query, DB = double-blind, KM = Kaplan-Meier approach, OL = open-label, SAE = serious adverse event, SMQ = standardized MedDRA query.

# 8 DEFINITION OF SUBGROUPS

Not Applicable

<sup>\*</sup>AEs of special interest includes: liver abnormalities, anemia/ hemoglobin decrease, edema, hypotension.

## 9 GENERAL STATISTICAL METHODOLOGY

# 9.1 Overall testing strategy

Not Applicable

# 9.2 General rules for data presentations

Data will be listed by country, site and DB treatment group and OL overall. Data will be summarized by appropriate descriptive statistics:

- Number of non-missing observations, mean, standard deviation, minimum, median and maximum for continuous variables.
- Number of events, number of censored observations and Kaplan-Meier estimates of the survival function for time-to-event variables.
- Number of non-missing observations, number of missing observations and frequency with percentage per category for categorical variables.
- Absolute changes from baseline are defined as: post-baseline value minus baseline value, i.e., a positive sign indicates an increase as compared to baseline.
- A percentage (relative) change from baseline is defined as the absolute change from baseline divided by the baseline value (if the baseline value is > 0) and then multiplied by 100.

Data will be presented for cohorts defined in section 2.1 (Table 2).

# 9.3 Display of patients disposition, protocol deviations and analysis set

## 9.3.1 Subject disposition

The number of patients included in each cohort will be summarized by treatment received in DB/OL.

The number and percentage of patients in analysis populations will be reported per cohort: Macitentan 10 mg (DB/OL) cohort broken down by treatment received in OL (10 mg/None, 10 mg/10 mg) and overall, and Macitentan 10 mg (OL) broken down by DB randomization groups (Placebo/ 10 mg, 3 mg/10 mg, 10 mg/10 mg) and overall.

Patients who completed study treatment as per protocol, who prematurely discontinued study drug as well as the reason for study drug discontinuation, will be reported the same way.

The coded reasons (Actelion Study Drug Log dictionary) are displayed in the summary.

Additionally, study drug discontinuation rates adjusted on person-year of study duration will be summarized with associated 95% CL as detailed in section 10.4.


#### 9.3.2 Protocol deviations

Protocol deviations will be reported as per Appendix E for the Macitentan 10 mg OL cohort.

PDs classified as "Important PD" will be summarized with a frequency table for SERAPHIN OL, the table should have columns corresponding to DB treatment group and total.

A listing of all protocol deviations in OL will be provided with a flag indicating whether the deviation is "Important PD".

A separate listing of all protocol deviations related to Covid-19 will be provided.

# 9.4 Analyses of patient characteristics

## 9.4.1 Demographics

For each cohort, demographics will be summarized descriptively. Macitentan 10 mg OL will be summarized Overall and per initial randomized treatment group.

#### 9.4.2 Baseline disease characteristics

For each cohort baseline disease characteristics will be summarized descriptively. Macitentan 10 mg OL will be summarized overall and by initial randomized treatment arm.

## 9.4.3 Other baseline characteristics

For each cohort other baseline characteristics will be summarized descriptively. Macitentan 10 mg OL will be summarized overall and per initial randomized treatment group.

## 9.4.4 Medical history

Medical history will not be summarized for this CSR.

### 9.4.5 Previous and concomitant medications

For study reporting purposes, all therapies collected in the AC-055-303 (SERAPHIN OL) CRF page 105 will be reported in the patient listings with the appropriate flags for previous/concomitant status, started before/after EOT.

Study-treatment concomitant therapies will be summarized by therapeutic organ class and PT.

A summary of concomitant PAH therapy at baseline (for baseline DB and separately baseline OL) will be summarizing the number and percentages of patients taking at least one PAH therapy, i.e. at least one PDE-5 inhibitor, at least one prostanoids and will be also summarized for each PT in these classifications as per section 5.2.5.2.

Concomitant medications will be summarized by each cohort, presenting the numbers of patients and associated percentages having any concomitant medication, by PT presented


by descending frequency of the total macitentan OL cohort PT incidence. Multiple medications (PT) taken by a single patient will only be counted once.

The following summaries will be presented for each cohort:

- A summary of concomitant PAH therapy at baseline (for baseline DB and separately baseline OL) including the number and percentages of patients taking
  - o at least one PAH therapy, i.e., at least one PDE-5 inhibitor, at least one prostanoid. Note: patients may receive more than one treatment and may be included in more than one treatment class.
- A summary of concomitant medication use at baseline of all medications taken by at least 5.0% patients in any cohort, by PT
- A summary of concomitant medication use during the study (at least 5.0% in any cohort), by PT.

A listing of concomitant medications will be provided.

# 9.5 Analysis of study treatment exposure and compliance

# 9.5.1 Exposure

Duration of treatment exposure for both cohorts, expressed in months, will be summarized descriptively. The distribution of exposure time by class intervals (in 6-month increments e.g., < 6 months, 6 - < 12 months, 84 - < 90 months, until the end of study) will be also tabulated to show the number and percentage of patients in each class interval. In addition, patient year exposure is displayed and is derived as the duration of exposure each patient received treatment in days, as defined above, divided by 365.25.

A listing of duration of Macitentan exposure and reasons for study drug discontinuation will be provided for the Macitentan 10 mg OL cohort (overall and by initial randomization).

## 9.5.2 Compliance with study treatment

Not applicable

# 9.6 Analysis of the exploratory efficacy variable(s)

### 9.6.1 Hypothesis and statistical model

Not applicable - the study is descriptive.


# 9.7 Analysis of safety variables

All safety analyses will be presented for Macitentan 10 mg OL overall and by randomization group, as well as for the Macitentan 10 mg DB/OL cohort.

All safety data will be included in listings, with flags for treatment-emergent and quantitative abnormalities, where appropriate (separately for initial randomization in DB groups).

#### 9.7.1 Adverse events

For all dosed patients all AEs captured from signature of informed will be reported in the patient listings.

A table presenting an overall summary of the proportion of patients with at least one treatment-emergent adverse event, one treatment-emergent AE of special interest, one treatment-emergent AE leading to treatment discontinuation, one treatment-emergent SAE, one treatment-emergent SAE with fatal outcome and the proportion of deaths will be provided.

Treatment-emergent AEs will be summarized by presenting the number and percentage of patients having any AE, having an AE in each primary system organ class (SOC), and having each individual AE (by PT) by descending PT frequency and separately by descending SOC/PT.

Exposure adjusted incidence rates will be also tabulated with two-sided 95% CLs (using method 1 and separately method 2).

Treatment-emergent AEs related to study drug will be summarized by presenting the number and percentage of patients having any AE, having an AE in each primary SOC, and having each individual AE (by PT) by descending PT frequency and separately by descending SOC/PT.

Treatment-emergent AEs will be also summarized by worst intensity by presenting the number and percentage of patients having any AE, having an AE in each primary SOC, and having each individual AE (by PT) by descending PT frequency and separately by descending SOC/PT.

### 9.7.2 Deaths, other serious adverse events

### 9.7.2.1 Death

Data for deaths will be summarized for both cohorts as below.

The number and percentage of treatment-emergent deaths will be presented from study start up to EOT+28 days. The number of deaths after EOT+28 days will be presented separately. In addition a summary of all deaths up to the study closure will be summarized.


Cause of death will be tabulated by SOC (with patients counted once within each SOC), and separately by PT (with patients counted once for each PT). SOC and PT will be presented by descending frequency in the OL cohort.

Exposure adjusted incidence rates will be also tabulated with two-sided 95% CLs.

A listing of all deaths (i.e., treatment-emergent and non-treatment-emergent events) is provided. Treatment-emergent deaths are flagged.

#### 9.7.2.2 *Time to death*

An analysis for survival up to study closure will be done, with end of study defined on a study basis (i.e. the data cut corresponding to data base lock).

For both cohorts, the proportion of patients surviving will be estimated by the Kaplan-Meier (KM) product-limit method and summarized for each group at pre-specified time-points (i.e., Day 0/Baseline, Month 6, Month 12, etc.), presenting number of patients at risk, number of patients with event (%), number of patients censored (%), KM estimates, and two-sided 95% CLs for the KM estimates. The standard error of the KM estimate will be calculated using Greenwood's formula [Collett 1994].

KM plot for time to death will be provided and will be truncated at the time when less than 10% of the patients within the treatment group are still at risk [Pocock 2002] or up to 108 months timepoint, whichever comes later.

The median time to death will be estimated from the KM curves, with corresponding 25% and 75% percentiles and associated 95% confidence intervals using the method of Brookmeyer [Brookmeyer 1982].

The corresponding listing of time to death will be provided.

Summary of study follow-up time will be summarized.

Details regarding how time to death is calculated are given in Section 5. SAS code examples are given in Appendix F.

#### 9.7.2.3 Serious adverse events

The number and percentage of patients experiencing at least one serious TEAE will be presented by descending within each SOC /PT and separately descending PT frequency. Exposure adjusted incidence rates will be tabulated with two-sided 95% CLs.

The number and percentage of patients experiencing at least one SAE after study drug termination will be summarized separately.

A listing of all SAEs (i.e., treatment-emergent and non-treatment-emergent events) will be provided for each analysis set. Serious TEAEs are flagged.


# 9.7.2.4 Adverse events leading to study treatment discontinuations

Adverse events leading to study treatment discontinuation will be described similarly as the SAEs

# 9.7.2.5 Other significant adverse events

The number and percentage of patients experiencing at least one TEAE of special interest will be presented by descending PT frequency for each AE of special interest.

The summaries include the exposure-adjusted incidence rates with associated 95% CLs.

Patient listing of AEs of special interest will be provided.

# 9.7.3 Laboratory tests

Absolute values and change from baseline values of all laboratory parameters described in section 5.6.8.1 will be summarized by visit. Time windows of +/- 15 days will be used as per Table 7.

Table 7 Time windows for all assessments up to EOT+28 days

| Mapping of visits<br>LFTs: | Study day<br>(nominal value) | Lower Limit study day | Upper Limit study day |
|---|---|---|---|
| Month 1 | 30 | 2 | 45 |
| Month 2 | 60 | 46 | 75 |
| Month 3 | 90 | 76 | 105 |
| Month 4 | 120 | 106 | 135 |
| Month 5 | 150 | 136 | 165 |
| Month 6 | 180 | 166 | 195 |
| Month 7 | 210 | 196 | 225 |
| Month 8 | 240 | 226 | 255 |
| Month 9 | 270 | 256 | 285 |
| Month 10 | 300 | 286 | 315 |
| Month 11 | 330 | 316 | 345 |
| Month 12 | 360 | 346 | 375 |
| Month 13 | 390 | 376 | 405 |
| Month 14 | 420 | 406 | 435 |
| Month 15 | 450 | 436 | 465 |
| Month 16 | 480 | 466 | 495 |
| Month 17 | 510 | 496 | 525 |
| Month 18 | 540 | 526 | 555 |

| Mapping of visits LFTs: | Study day<br>(nominal value) | Lower Limit study day | Upper Limit study day |
|---|---|---|---|
| Month 19 | 570 | 556 | 585 |
| Month 20 | 600 | 586 | 615 |
| Month 21 | 630 | 616 | 645 |
| Month 22 | 660 | 646 | 675 |
| Month 23 | 690 | 676 | 705 |
| Month 24 | 720 | 706 | 735 |
| Month 25 | 750 | 736 | 765 |
| Month 26 | 780 | 766 | 795 |
| Month 27 | 810 | 796 | 825 |
| Month 28 | 840 | 826 | 855 |
| Month 29 | 870 | 856 | 885 |
| Month 30 | 900 | 886 | 915 |
| Month 31 | 930 | 916 | 945 |
| Month 32 | 960 | 946 | 975 |
| Month 33 | 990 | 976 | 1005 |
| Month 34 | 1020 | 1006 | 1035 |
| Month 35 | 1050 | 1036 | 1065 |
| Month 36 | 1080 | 1066 | 1095 |
| Month 37 | 1110 | 1096 | 1125 |
| Month 38 | 1140 | 1126 | 1155 |
| Month 39 | 1170 | 1156 | 1185 |
| Month 40 | 1200 | 1186 | 1215 |
| Month 41 | 1230 | 1216 | 1245 |
| Month X | X*30 | X*30<br>- 14 | X*30<br>+15 |
| Month 126 | 3780 | 3766 | 3795 |

Summary statistics of worst abnormalities post baseline will be provided for each parameter as described in Table 5 for Low abnormalities and high abnormalities separately.

A supportive listing of all laboratory data is provided with a flag for abnormal values.

## 9.7.4 Incidence of abnormal liver tests (including unscheduled visits)

Liver tests for ALT, AST, and total bilirubin will be presented using incidence (n [%]) with the two-sided 95% CLs based on Wald approximation, and tabulated for patients with abnormalities. Exposure adjusted incidence rates will be tabulated with two-sided 95% CLs.

A supportive listing will be provided for with all liver tests laboratory data collected. Treatment-emergent results will be flagged.

Using "evaluation of drug-induced serious hepatotoxicity" (eDISH) plots, graphical representations of total bilirubin versus ALT will be produced for each initial randomized treatment group and for Overall Macitentan 10 mg OL cohort to identify possible Hy's Law cases. The graph presents, for each patient, the peak total bilirubin  $\times$  ULN against the peak ALT  $\times$  ULN in the same reporting period, on a log10 scale. Two reference lines will be plotted identifying the 2  $\times$  ULN for total bilirubin and 3  $\times$  ULN for ALT. The peak is the maximum value from treatment start to last available assessment within the treatment period and up to EOT plus 28 days.

A supportive listing presents all liver test data over time for all patients in Hy's Law quadrant.

# 9.7.5 Incidence of abnormal hemoglobin values

Patient counts and percent (with corresponding two-sided 95% CLs based on the Wald method and using Poisson model with time as an offset variable) for the categories of Hgb abnormality occurring at any time post-baseline up to EOT + 28 days will be presented.

Exposure adjusted incidence will be tabulated with two-sided 95% CLs.

A supportive listing provides presents all hemoglobin values collected. Treatment-emergent results will be flagged.

### 9.7.6 Other laboratory parameters

All other laboratory parameters collected are listed.

## 10 GENERAL DEFINITIONS AND DERIVATIONS

### **10.1** Dates of interest

The dates of interest were defined in section "Definition of Variables".

# 10.2 Macitentan DB/OL treatment emergent period (for safety variables reporting)

The Macitentan DB/OL treatment-emergent period is defined as the period from the first intake of Macitentan to the Macitentan EOT date (max[EOT302, EOT303]) + 28 days.

For laboratory analyses, the Macitentan DB/OL treatment-emergent period defined above starts from the first administration of Macitentan.

# 10.3 Macitentan OL treatment emergent period (for safety variables reporting)

The Macitentan OL treatment-emergent period is defined as the period from **STRT303** up to the EOT303 + 28 days.

For laboratory analyses, the Macitentan OL treatment-emergent period defined above starts from Macitentan start date in OL.

# 10.4 Adjusted incidence rates

In order to account for differences in the duration of exposure of study treatment among the patient cohorts, incidence rates of AEs, SAEs, AEs leading to discontinuation, AESI, and deaths will be presented as adjusted for patient-years exposure (PYE).

There will be two slightly different methods:

Method 1: The same approach as in the original NDA submission in 2012 will be applied [D-12.548], where total treatment exposure for each patient is included in the calculation. This will be applied in order to make comparison versus the original submission.

Person-time will be calculated by summing the days of treatment duration (" EOT-STRT302 +1 OR EOT-STRT303 +1 as per section 5.3) for each patient.

PYE will be calculated by dividing the total patient time by 365.25 days.

The incidence rate for an AE per 100 person-years will be calculated by dividing the number of patients with AEs by the PYE and multiplying by 100.

Adjusted Incidence Rate = 100 x (Number of patients with at least one AE/PYE)

### Method 2:

A similar approach as in the original NDA submission in 2012 but the treatment exposure will be calculated up to the first event for patients with events [Siddiqui 2009]. The same as in the Method 1 except:

Person-time will be calculated:

i) by summing the days of treatment duration (EOT- STRT303 +1 as per section 5.3.1) for patients without events,


- ii) by summing the days of treatment duration up to the start date of first event (min[date of first event, EOT] STRT303] + 1) for patients with event,
- iii) all other calculations for adjusted incidence rate follow the Method-1.

The adjusted incidence rate will be interpreted as the number of events occurring in 100-patient years. It is based on the assumption that the occurrences of a specific event are following an independent Poisson process, so the events occur with a constant rate over time. Hence, for each treatment group, the 95% Confidence Limit (CL) of the adjusted incidence rate will be computed using a Poisson regression model with log of time at risk as an offset (SAS PROC GENMOD, see Appendix B for code example).

Note for programming: For AEs, SAEs, AEs leading to discontinuation, AESI group level, and deaths, the overall adjusted event rates will be presented using method 1 (i.e. adjusted rate will not be presented for each PT, except for AEs, where will be presented overall and by SOC). Method 2 will be applied only for AEs and AESI group level.

## 11 HANDLING OF MISSING/INCOMPLETE DATE AND TIME FIELDS

The missing or incomplete dates for the variables defined below will be derived as follows:

- 1. Dates will be split into 3 parts: year, month and day. Year is the top-level, month is medium level and day is low-level. If a part expected to contain a number is numeric but the value is outside a valid range, the complete date is handled as missing. For example, if date = 44Nov2000 the whole date is considered to be missing.
- 2. If a part expected to contain a number is not numeric, i.e., contains values such as for example ND, NA, --, ??, 2?, it is considered as missing.
- 3. If a part is missing, all other parts of a lower level are considered to be missing. This means that a ddmmyy date '21ND99' is considered as '---99'.
- 4. Missing parts are changed into acceptable non-missing values in a way depending on the type of date to be replaced.

'lower limit' and 'upper limit' refer to the minimum or maximum, respectively, of a possible date. For example, if the day is missing, the lowest limit is the first day of the given month and the upper limit is the last day of the given month. If the day and month are missing, the lower limit refers to the first day of the given year and the upper limit to the last day of the given year. The earliest and the latest of different dates refer to the first or last date, respectively, when ordered in sequence. All other missing or incomplete data not mentioned below are treated as missing.

| Type of date/time | Date/time is incomplete | Date/time is missing |
|---|---|---|
| Date of birth | Day missing: 15th of the month | No replacement |
| | Day and month missing: 30th of June | |
| Type of date/time | Date/time is incomplete | Date/time is missing |
|---|---|---|
| EOT302 | <ul> <li>Use the earliest date between the:</li> <li>upper limit</li> <li>last contact date (LCTC)</li> <li>date of death (if applicable)</li> <li>treatment start date of 303-1</li> </ul> | Use the earliest date between the: • 6 months after last available dispensing visit date, i.e., 180 days + randomization or Month 6 or Month 12 or Month 18, visit date • last contact date (LCTC) • date of death (if applicable) • Start treatment date of 303-1 |
| ЕОТ303 | <ul> <li>Use the earliest date between the:</li> <li>upper limit</li> <li>last contact date (LCTC)</li> <li>date of death (if applicable)</li> </ul> | <ul><li>Use the earliest date between</li><li>the:</li><li>last contact date (LCTC)</li><li>date of death (if applicable)</li></ul> |
| DOD - Date of death | Use the lower limit if day is missing | |
| EOS303 | <ul><li>Use the earliest date between the:</li><li>upper limit</li><li>date of death (if applicable)</li></ul> | |
| AE resolution date | The upper limit | No approximation, the AE is considered as ongoing. |

| Type of date/time | Date/time is incomplete | Date/time is missing |
|---|---|---|
| AE onset date | If the end date of the AE is not before the start of study treatment, and if the study treatment start falls in the range of possible dates, it is the study treatment start date. In all other cases, it is the lower limit. Of note, treatment start date is STRT302 for Macitentan 3 mg or 10 mg (DB/OL) and STRT303 for Macitentan 10 mg (OL). | The earlier of the end date of the AE and the start of study treatment (STRT302 for Macitentan 3 mg or 10 mg [DB/OL] and STRT303 for macitentan 10 mg [OL]). |
| Previous/ | Lower limit except when: | No replacement, the |
| concomitant | Not tagged as ongoing at baseline | medication is considered to |
| medication | AND | have started before the study |
| start date | Medication stop date not collected or with the upper limit after study drug start | |
| | AND | |
| | The treatment start day falls in the range of possible dates. | |
| | In which case it is the study drug start day | |
| Previous/ | Note that Medication stop date will not | No replacement |
| concomitant | be imputed; however the upper limit may be used in determining the | |
| medication | medication start date derivation. | |
| end date | | |


| Type of date/time | Date/time is incomplete | Date/time is missing |
|---|---|---|
| AE resolution time | Time partially entered not allowed (considered as missing) | Taken as "23:59" if the corresponding AE resolution date is not missing, otherwise no replacement |

#### Notes:

- Patient PPD in Macitentan 10 mg (DB/OL) group was considered as having no PAH therapy at baseline in analysis of DB data in 2012, based on a rule that if the end date was partial and upper limit of that end date was after the study drug start date and the tick box ongoing at baseline was not ticked the medication was ended before the study start date. This patient has a record of Sildenafil with a start date of PPD and and an end date of PPD and a study drug start date of PPD and a study drug start date is after the study drug start date. This medication is considered as ongoing at baseline.
- Patient PPD in Macitentan 3 mg (DB/OL) group (Macitentan start date PPD ) was considered as having no PAH therapy at baseline in analysis of DB data in 2012 (SILDENAFIL/ Start date=PPD '/ End Date=PPD '/

## 12 LIST OF SUMMARY TABLES, LISTINGS AND FIGURES

## 12.1 Patients disposition

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 1 | T | Number of Patients in the different patient cohorts | SAF |
| Table 2 | Т | Number of Patients in the different<br>patient cohorts and Reasons for<br>Study Drug Discontinuation | SAF |

T=Summary table, L= Listing, F=Figure

#### 12.2 Protocol deviations

| Output<br>name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 3 | T | Summary of Important protocol deviations. | Macitentan<br>10 mg OL |
| Listing 1 | L | All protocol deviations | Macitentan<br>10 mg OL |
| Listing 1.1 | L | Protocol deviations related to Covid-19 | Macitentan<br>10 mg OL |

## 12.3 Patients characteristics

## 12.3.1 Demographics and Patient Characteristics

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 4 | T | Summary of Demographic and Patient Characteristics | SAF |

## 12.3.2 Previous and concomitant therapies

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 5 | Т | Summary of concomitant PAH therapy (for baseline DB and separately baseline OL) | SAF |
| Table 6 | Т | Summary of concomitant medication use at baseline (at least 5% in any cohort), by preferred term | SAF |
| Table 7 | T | Summary of concomitant medication use during the study (at least 5% in any cohort), by preferred term | SAF |
| Listing 2 | L | Patient listing of concomitant medications | SAF |
| Listing 3 | L | Discrepancies in previous and concomitant medications | SAF |

# 12.4 Study treatment exposure and compliance

## 12.4.1 Exposure

| Output<br>name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 8 | Т | Summary of duration of Exposure to Study Drug | SAF |
| Listing 4 | L | Patient listing of exposure and reasons for study drug discontinuation | SAF |

# 12.5 Safety analyses

## 12.5.1 Adverse events

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 9 | T | Proportion of patients with AEs, AEs of special interest, SAEs, SAEs with fatal outcome, AEs leading to permanent study drug discontinuation and number of patients who died from treatment start up to EOT+28 days | SAF |
| Table 10 | T | Proportion of patients with AEs occurring from treatment start up to EOT+28 days by PT | SAF |
| Table 11 | T | Proportion of patients with AEs occurring from treatment start up to EOT+28 days by SOC and by PT | SAF |
| Table 12 | T | Proportion of patients with AEs related to study drug occurring from treatment start up to EOT+28 days by PT | SAF |
| Table 13 | T | Proportion of patients with AEs related to study drug occurring from treatment start up to EOT+28 days by SOC and by PT | SAF |
| Table 14 | T | Proportion of patients with AEs by<br>severity occurring from treatment<br>start up to EOT+28 days by PT | SAF |
| Table 15 | T | Proportion of patients with AEs by<br>severity occurring from treatment<br>start up to EOT+28 days by SOC and<br>by PT | SAF |
| Listing 5 | L | Patient listing of all adverse events | SAF |


## **12.5.2 Deaths**

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 16 | T | Deaths occurring from treatment start<br>up to EOT+28 days by cause (by<br>SOC and by PT) | SAF |
| Table 17 | T | Deaths occurring from treatment start up to EOT+28 days by cause (by PT) | SAF |
| Table 18 | T | Deaths occurring after EOT+28 days (by PT) | SAF |
| Table 19 | T | Deaths occurring after EOT+28 days (by SOC and by PT) | SAF |
| Table 20 | T | Deaths occurring from treatment start<br>up to the study closure by cause (by<br>PT) | SAF |
| Table 21 | T | Deaths occurring from treatment start<br>up to the study closure by cause (by<br>SOC and by PT) | SAF |
| Listing 6 | L | All deaths | SAF |

## 12.5.3 Time to death

| Output<br>name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 22 | T | Summary of Time to Death up to the study closure | SAF |
| Listing 7 | L | Patient listing of time to deaths up to study closure | SAF |
| Table 23 | T | Summary of study follow up time - reverse Kaplan Meier method | SAF |
| Figure 1.1 | F | Kaplan Meier curve of Time to<br>Death up to the study closure | Macitentan<br>10 mg<br>(DB/OL) |
| Figure 1.2 | F | Kaplan Meier curve of Time to<br>Death up to the study closure | Macitentan<br>10 mg (OL) |

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Figure 1.3 | F | Kaplan Meier curve of Time to<br>Death up to the study closure by<br>randomization group. | |

## 12.5.4 Serious adverse events

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 24 | T | Proportion of patients with SAEs occurring from treatment start up to EOT+28 days by PT | SAF |
| Table 25 | T | Proportion of patients with SAEs occurring from treatment start up to EOT+28 days by SOC and by PT | SAF |
| Table 26 | T | Proportion of patients with SAEs occurring after study drug termination by PT | SAF |
| Table 27 | T | Proportion of patients with SAEs occurring after study drug termination by SOC and by PT | SAF |
| Listing 8 | L | Patient listing of all SAEs | SAF |

## 12.5.5 Adverse events leading to treatment discontinuation

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 28 | T | Proportion of patients with<br>treatment-emergent adverse events<br>leading to permanent study drug<br>discontinuation by PT | SAF |
| Table 29 | Т | Proportion of patients with<br>treatment-emergent adverse events<br>leading to permanent study drug<br>discontinuation by SOC and by PT | SAF |


| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Listing 9 | L | Treatment-emergent adverse events leading to permanent study drug discontinuation | SAF |

## 12.5.6 Other significant adverse events

| Output name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 30 | T | Proportion of Patients with AEs of special interest occurring from treatment start up to EOT+28 days by PT: <smq x=""></smq> | SAF |
| Listing<br>10 | L | Averse events of special interest <smq x=""></smq> | SAF |

## 12.6 **Laboratory tests**

| Output<br>name | Display | Title (Description) | Analysis set(s) |
|---|---|---|---|
| Table 31 | T | Summary of absolute and absolute change for laboratory parameters from Macitentan 10 mg DB baseline, by analysis visit - Macitentan 10 mg (DB/OL) | SAF |
| Table 32 | T | Summary of absolute and absolute change for laboratory parameters from Macitentan 10 mg OL baseline, by analysis visit - Macitentan 10 mg (OL) | SAF |
| Table 33 | T | Proportion of patients with incidence of all laboratory abnormalities occurring from treatment start up to EOT+28 days | SAF |
| Table 34 | T | Proportion of patients with Liver tests Abnormalities occurring from treatment start up to EOT+28 days | SAF |
| Listing 11 | L | Abnormal Liver tests (ALT or<br>AST > 3 x ULN) or total bilirubin ><br>2 x ULN | SAF |


Listing 15 L

SAF


#### Figure 2 F Peak Total Bilirubin vs. peak ALT SAF (eDish plot) (one per cohort) Listing 12 L Patient listing of liver test data for all SAF patients in Hy's Law quadrant over time. Table 35 T Proportion of patients with incidence SAF of hemoglobin abnormalities occurring from treatment start up to EOT+28 days Listing 13 L Hemoglobin abnormalities (Hgb ≤ SAF 100 g/LListing 14 L Patient listing of all other SAF abnormalities

Patient listing of all laboratory data


#### 13 REFERENCES

- [D-12.425] A multicenter, double-blind, randomized, placebo controlled, parallel group, event driven, Phase III study to assess the effects of macitentan on morbidity and mortality in patients with symptomatic pulmonary arterial hypertension. Actelion Pharmaceuticals Ltd; Final Study Report AC-055-302, 31 August 2012. Previously submitted to NDA 204410, sequence 0000 on 19 October 2012, Module 5.3.5.1.
- [D-12.548] Statistical Analysis Plan for Integrated Safety Analysis. Actelion Pharmaceuticals Ltd; 31 August 2012. Previously submitted to NDA 204410, sequence 0000 on 19 October 2012, Module 5.3.5.3, Appendix 1A.
- [Brookmeyer 1982] Brookmeyer R, Crowley JA. CI for the median survival time. Biometrics. 1982; 38:29-41.
- [Collett 1994] Collett D. Modelling survival data in medical research. London: Chapman & Hall; 1994.
- [Holden 2003] Holden WL, Juhaeri J, Dai W. Benefit-risk analysis: a proposal using quantitative methods. Pharmacoepidemiol Drug Saf. 2003; 2:611-6.
- [Pocock 2002] Pocock SJ, Clayton TC, Altman DG. Survival plots of time-to-event outcomes in clinical trials: good practice and pitfalls. The Lancet 2002;359:1686-89.
- [Siddiqui 2009]. Siddiqui O. Statistical Methods to Analyze Adverse Events Data of Randomized Clinical Trials. Journal of Biopharmaceutical Statistics. 2009;19(5): 889-899.
- [Ware 2000] Ware JE, Kosinski M, Dewey JE. How to Score Version Two of the SF-36 Health Survey. Lincoln, RI: QualityMetric, Incorporated, 2000.

## 14 APPENDICES

## Appendix A Protocol Synopsis AC-055-303 (SERAPHIN OL)

| TITLE | Long-term single-arm open-label extension study of the SERAPHIN study, to assess the safety and tolerability of macitentan/ACT-064992 in patients with symptomatic pulmonary arterial hypertension. | | | | | |
|---|---|---|---|---|---|---|
| ACRONYM | | | with an <u>ERA</u> inve cli <u>N</u> ical outc | | | |
| OBJECTIVES | To assess the long-term safety and tolerability of ACT-064992 in patients with symptomatic pulmonary arterial hypertension (PAH). | | | | | |
| DESIGN / PHASE | Multicenter, o | pen-label | (OL) extension | n, single- | arm, Phase III s | study |
| STUDY PLANNED<br>DURATION | First patient<br>First visit | Q4/07 | Last patient<br>First visit | Q1/12 | Last patient<br>Last visit | Open |
| CENTERS<br>/ COUNTRIES | Approximately 180 centers in about 40 countries. | | | | | |
| PATIENTS / GROUPS | Up to 699 patients in one group. | | | | | |
| INCLUSION CRITERIA | <ul> <li>Signed informed consent prior to initiation of any study-mandated procedure.</li> <li>Patients with pulmonary arterial hypertension and having completed the event-driven study, AC-055-302/SERAPHIN, or</li> </ul> | | | | | |
| | Patients who have experienced a clinical worsening of PAF AC-055-302/SERAPHIN and for whom a written approva roll over into this study has been obtained from the Sponsor. | | oval to | | | |
| Women of childbearing potential must have a treatment serum pregnancy test and must use a re of contraception during study treatment and for at after study treatment termination. | | use a reliable | method | | | |


|------------------------------|

| EXCLUSION CRITERIA | Any major violation of protocol AC-055-302/SERAPHIN. |
|---|---|
| | Pregnancy or breast-feeding. |
| | • AST and/or ALT > 3 times the upper limit of the normal range. |
| | <ul> <li>Any known factor or disease that might interfere with treatment<br/>compliance, study conduct or interpretation of the results, such as<br/>drug or alcohol dependence or psychiatric disease.</li> </ul> |
| | • Known hypersensitivity to ACT-064992 or any of the excipients. |

## Appendix B Example SAS code for incidence rates and 95% CL

Note: time should be in years for GENMOD

```
** example code to show derivation of rate and CI based on dummy data **;
** Create dummy data **;
data aA:
 tot eve=0;
 tot time=0;
 do pn=1 to 110:
  time=ranuni(546546)*1000; ** time to event**;
  eve=(ranuni(5454)<.10); ** event or censor **;
  tot eve+eve;
  tot time+time;
  1 time=log(time/365.25);
  if pn=110 then do;
   incidence=100*tot eve/(tot time/365.25); **incidence rate **;
  end:
  output;
 end;
run;
proc genmod data=aa;
 model eve= / dist=poisson link=log offset=1 time; /*** here is the exposure time in offset***/
 output out=out p=pcount xbeta=xb stdxbeta=std;
 ods output ParameterEstimates=param;
run;
data predrates;
 set out;
 obsrate=eve/time;
                       /* observed rate */
 lograte=xb-l time;
 prate=100*exp(lograte); /* predicted rate */
 lcl=100*exp(lograte-probit(.975)*std); ** Lower Limit **;
 ucl=100*exp(lograte+probit(.975)*std); ** upper Limit **;
run;
** derivation also available in PARAM**;
data param2;
 set param(WHERE=(parameter=("Intercept")));
 prate=100*exp(estimate);
 lcl=100*exp(LowerWaldCL);
 ucl=100*exp(UpperWaldCL);
run;
```


Statistical Analysis Plan EDMS-RIM-297091

## Appendix C Definition of AEs of special interest

#### 1 LIVER ABNORMALITIES

AEs are included in this grouping if they contain an event PT within the 'Hepatic disorders' SMQ, including all of its sub-SMQs, with the exception of the 'Liver-related coagulation and bleeding disturbances' sub-SMQ and the PTs 'Ascites', 'Bacterascites', 'Biliary ascites', and 'Haemorrhagic ascites', i.e., any of the following MedDRA PTs:

5'nucleotidase increased

Accessory liver lobe

Acquired hepatocerebral degeneration

Acute fatty liver of pregnancy

Acute graft versus host disease in liver

Acute hepatic failure

Acute hepatitis B

Acute hepatitis C

Acute on chronic liver failure

Acute yellow liver atrophy

Adenoviral hepatitis

Alagille syndrome

Alanine aminotransferase abnormal

Alanine aminotransferase increased

Alcoholic liver disease

Allergic hepatitis

Alloimmune hepatitis

Ammonia abnormal

Ammonia increased

Anorectal varices

Anorectal varices haemorrhage

Aspartate aminotransferase abnormal

Aspartate aminotransferase increased

AST/ALT ratio abnormal

Asterixis

\_

<sup>&</sup>lt;sup>1</sup> Excluded PTs: Ascites, Bacterascites, Biliary ascites, Haemorrhagic ascites, Acquired factor IX deficiency, Acquired factor VIII deficiency, Acquired factor XI deficiency, Acquired antithrombin III deficiency, Acquired protein S deficiency, Anti factor X activity abnormal, Anti factor X activity decreased, Anti factor X activity increased, Antithrombin III decreased, Blood fibrinogen abnormal, Blood fibrinogen decreased, Blood thrombin abnormal, Blood thromboplastin decreased, Coagulation factor decreased, Coagulation factor IX level abnormal, Coagulation factor V level abnormal, Coagulation factor V level decreased, Coagulation factor VIII level abnormal, Coagulation factor X level decreased, Hyperfibrinolysis, Hypocoagulable state, Hypofibrinogenaemia, Hypoprothrombinaemia, Hypothrombinaemia, Hypothromboplastinaemia, International normalised ratio abnormal, International normalised ratio increased, Protein C decreased, Protein S abnormal, Protein S decreased, Prothrombin time ratio abnormal, Prothrombin time prolonged.


Statistical Analysis Plan EDMS-RIM-297091

Asymptomatic viral hepatitis

Autoimmune hepatitis

Benign hepatic neoplasm

Benign hepatobiliary neoplasm

Bile output abnormal

Bile output decreased

Biliary cirrhosis

Biliary fibrosis

Bilirubin conjugated abnormal

Bilirubin conjugated increased

Bilirubin excretion disorder

Bilirubin urine present

Biopsy liver abnormal

Blood alkaline phosphatase abnormal

Blood alkaline phosphatase increased

Blood bilirubin abnormal

Blood bilirubin increased

Blood bilirubin unconjugated increased

Blood cholinesterase abnormal

Blood cholinesterase decreased

Bromosulphthalein test abnormal

Cardiohepatic syndrome

Cerebrohepatorenal syndrome

Child-Pugh-Turcotte score abnormal

Child-Pugh-Turcotte score increased

Cholaemia

Cholangiosarcoma

Cholestasis

Cholestasis of pregnancy

Cholestatic liver injury

Cholestatic pruritus

Chronic graft versus host disease in liver

Chronic hepatic failure

Chronic hepatitis

Chronic hepatitis B

Chronic hepatitis C

Cirrhosis alcoholic

Coma hepatic

Complications of transplanted liver

Computerised tomogram liver abnormal

Congenital absence of bile ducts

Congenital cystic disease of liver

Congenital hepatic fibrosis

Congenital hepatitis B infection

Congenital hepatobiliary anomaly


Statistical Analysis Plan EDMS-RIM-297091

#### Congenital hepatomegaly

Cryptogenic cirrhosis

Cystic fibrosis hepatic disease

Cytomegalovirus hepatitis

Deficiency of bile secretion

Diabetic hepatopathy

Dilatation intrahepatic duct congenital

Drug-induced liver injury

Duodenal varices

Fatty liver alcoholic

Focal nodular hyperplasia

Foetor hepaticus

Galactose elimination capacity test abnormal

Galactose elimination capacity test decreased

Gallbladder varices

Gamma-glutamyltransferase abnormal

Gamma-glutamyltransferase increased

Gastric variceal injection

Gastric variceal ligation

Gastric varices

Gastric varices haemorrhage

Gastrooesophageal variceal haemorrhage prophylaxis

Gianotti-Crosti syndrome

Glutamate dehydrogenase increased

Glycocholic acid increased

Glycogen storage disease type I

Glycogen storage disease type III

Glycogen storage disease type IV

Glycogen storage disease type VI

Graft versus host disease in liver

Granulomatous liver disease

Guanase increased

Haemangioma of liver

Haemorrhagic hepatic cyst

HBV-DNA polymerase increased

Hepaplastin abnormal

Hepaplastin decreased

Hepatectomy

Hepatic adenoma

Hepatic amoebiasis

Hepatic angiosarcoma

Hepatic artery flow decreased

Hepatic atrophy

Hepatic calcification

Hepatic cancer


#### Hepatic cancer metastatic

Hepatic cancer recurrent

Hepatic cancer stage I

Hepatic cancer stage II

Hepatic cancer stage III

Hepatic cancer stage IV

Hepatic candidiasis

Hepatic cirrhosis

Hepatic congestion

Hepatic cyst

Hepatic cyst infection

Hepatic cyst ruptured

Hepatic echinococciasis

Hepatic encephalopathy

Hepatic encephalopathy prophylaxis

Hepatic enzyme abnormal

Hepatic enzyme decreased

Hepatic enzyme increased

Hepatic failure

Hepatic fibrosis

Hepatic fibrosis marker abnormal

Hepatic fibrosis marker increased

Hepatic function abnormal

Hepatic gas gangrene

Hepatic haemangioma rupture

Hepatic hamartoma

Hepatic hydrothorax

Hepatic hypertrophy

Hepatic infection

Hepatic infection bacterial

Hepatic infection fungal

Hepatic infection helminthic

Hepatic infiltration eosinophilic

Hepatic lesion

Hepatic lymphocytic infiltration

Hepatic mass

Hepatic necrosis

Hepatic neoplasm

Hepatic pain

Hepatic sequestration

Hepatic steato-fibrosis

Hepatic steatosis

Hepatic vascular resistance increased

Hepatic venous pressure gradient abnormal

Hepatic venous pressure gradient increased


Hepatitis

Hepatitis A

Hepatitis A antibody abnormal

Hepatitis A antibody positive

Hepatitis A antigen positive

Hepatitis A virus test positive

Hepatitis acute

Hepatitis alcoholic

Hepatitis B

Hepatitis B antibody abnormal

Hepatitis B antibody positive

Hepatitis B core antibody positive

Hepatitis B core antigen positive

Hepatitis B DNA assay positive

Hepatitis B DNA increased

Hepatitis B e antibody positive

Hepatitis B e antigen positive

Hepatitis B reactivation

Hepatitis B surface antibody positive

Hepatitis B surface antigen positive

Hepatitis B virus test positive

Hepatitis C

Hepatitis C antibody positive

Hepatitis C core antibody positive

Hepatitis C RNA increased

Hepatitis C RNA positive

Hepatitis C virus test positive

Hepatitis cholestatic

Hepatitis chronic active

Hepatitis chronic persistent

Hepatitis D

Hepatitis D antibody positive

Hepatitis D antigen positive

Hepatitis D RNA positive

Hepatitis D virus test positive

Hepatitis E

Hepatitis E antibody abnormal

Hepatitis E antibody positive

Hepatitis E antigen positive

Hepatitis E virus test positive

Hepatitis F

Hepatitis fulminant

Hepatitis G

Hepatitis H

Hepatitis infectious mononucleosis


Statistical Analysis Plan EDMS-RIM-297091

Hepatitis mumps

Hepatitis neonatal

Hepatitis non-A non-B

Hepatitis non-A non-B non-C

Hepatitis post transfusion

Hepatitis syphilitic

Hepatitis toxic

Hepatitis toxoplasmal

Hepatitis viral

Hepatitis viral test positive

Hepatobiliary cancer

Hepatobiliary cancer in situ

Hepatobiliary cyst

Hepatobiliary disease

Hepatobiliary infection

Hepatobiliary neoplasm

Hepatobiliary scan abnormal

Hepatoblastoma

Hepatoblastoma recurrent

Hepatocellular carcinoma

Hepatocellular damage neonatal

Hepatocellular foamy cell syndrome

Hepatocellular injury

Hepato-lenticular degeneration

Hepatomegaly

Hepatopulmonary syndrome

Hepatorenal failure

Hepatorenal syndrome

Hepatosplenic abscess

Hepatosplenic candidiasis

Hepatosplenomegaly

Hepatosplenomegaly neonatal

Hepatotoxicity

Hereditary haemochromatosis

Herpes simplex hepatitis

Hyperammonaemia

Hyperbilirubinaemia

Hyperbilirubinaemia neonatal

Hypercholia

Hypertransaminasaemia

Hypoalbuminaemia

Icterus index increased

Immune-mediated hepatitis

Increased liver stiffness

Intestinal varices


Statistical Analysis Plan EDMS-RIM-297091

Intestinal varices haemorrhage

Intrahepatic portal hepatic venous fistula

Ischaemic hepatitis

Jaundice

Jaundice cholestatic

Jaundice hepatocellular

Jaundice neonatal

Kayser-Fleischer ring

Kernicterus

Leucine aminopeptidase increased

Liver ablation

Liver abscess

Liver and pancreas transplant rejection

Liver carcinoma ruptured

Liver dialysis

Liver disorder

Liver function test abnormal

Liver function test decreased

Liver function test increased

Liver induration

Liver injury

Liver iron concentration abnormal

Liver iron concentration increased

Liver operation

Liver palpable

Liver sarcoidosis

Liver scan abnormal

Liver tenderness

Liver transplant

Liver transplant failure

Liver transplant rejection

Lupoid hepatic cirrhosis

Lupus hepatitis

Magnetic resonance imaging liver abnormal

Magnetic resonance proton density fat fraction

measurement

Minimal hepatic encephalopathy

Mitochondrial aspartate aminotransferase increased

Mixed hepatocellular cholangiocarcinoma

Mixed liver injury

Model for end stage liver disease score abnormal

Model for end stage liver disease score increased

Molar ratio of total branched-chain amino acid to tyrosine

Multivisceral transplantation

Neonatal cholestasis


Statistical Analysis Plan EDMS-RIM-297091

Neonatal hepatomegaly

Nodular regenerative hyperplasia

Nonalcoholic fatty liver disease

Non-alcoholic steatohepatitis

Non-cirrhotic portal hypertension

Ocular icterus

Oedema due to hepatic disease

Oesophageal varices haemorrhage

Parenteral nutrition associated liver disease

Partial splenic embolisation

Perihepatic discomfort

Perinatal HBV infection

Peripancreatic varices

Periportal oedema

Peritoneal fluid protein abnormal

Peritoneal fluid protein decreased

Peritoneal fluid protein increased

Peritoneovenous shunt

Pneumobilia

Polycystic liver disease

Porphyria acute

Porphyria non-acute

Portal fibrosis

Portal hypertension

Portal hypertensive colopathy

Portal hypertensive enteropathy

Portal hypertensive gastropathy

Portal pyaemia

Portal shunt

Portal shunt procedure

Portal tract inflammation

Portal vein cavernous transformation

Portal vein dilatation

Portal vein flow decreased

Portal vein pressure increased

Portal venous system anomaly

Portopulmonary hypertension

Primary biliary cholangitis

Progressive familial intrahepatic cholestasis

Radiation hepatitis

Regenerative siderotic hepatic nodule

Renal and liver transplant

Retinol binding protein decreased

Retrograde portal vein flow

Reye's syndrome


Statistical Analysis Plan EDMS-RIM-297091

Reynold's syndrome

Schistosomiasis liver

Small-for-size liver syndrome

Spider naevus

Splenic varices

Splenic varices haemorrhage

Splenorenal shunt

Splenorenal shunt procedure

Spontaneous intrahepatic portosystemic venous shunt

Steatohepatitis

Stomal varices

Subacute hepatic failure

Sugiura procedure

Sustained viral response

Total bile acids increased

Transaminases abnormal

Transaminases increased

Ultrasound liver abnormal

Urine bilirubin increased

Urobilinogen urine decreased

Urobilinogen urine increased

Varices oesophageal

Varicose veins of abdominal wall

Viral hepatitis carrier

Weil's disease

White nipple sign

Withdrawal hepatitis

X-ray hepatobiliary abnormal

Yellow skin

Zieve syndrome

#### 2 EDEMA

AEs are included in this grouping if they contain an event with the MedDRA Preferred Term "Pulmonary congestion" or if within the SMQ "Haemodynamic oedema, effusions and fluid overload (SMQ)" with the exception of PTs containing "site", ie the case will be included if it contains an event with any of the following MedDRA PTs:

Acute pulmonary oedema

Amyloid related imaging abnormalities

Amyloid related imaging abnormality-microhaemorrhages and haemosiderin

Amyloid related imaging abnormality-oedema/effusion

Ascites

Bone marrow oedema


#### Bone marrow oedema syndrome

Bone swelling

Brain oedema

Bronchial oedema

Capillary leak syndrome

Cerebral oedema management

Cervix oedema

Circumoral swelling

Compression garment application

Cytotoxic oedema

Durotomy procedure

Effusion

Elephantiasis nostras verrucosa

Extensive swelling of vaccinated limb

Fluid overload

Fluid retention

Gallbladder oedema

Gastrointestinal oedema

Generalised oedema

Gestational oedema

Gravitational oedema

Heat oedema

Hydraemia

Hydrothorax

Hydrovarium

Hypervolaemia

Hypoosmolar state

Joint effusion

Joint swelling

Lipoedema

Localised oedema

Lymphoedema

Modified Rodnan skin score abnormal

Mouth swelling

Muscle oedema

Muscle swelling

Myocardial oedema

Negative pressure pulmonary oedema

Non-cardiogenic pulmonary oedema

Oedema

Oedema blister

Oedema due to cardiac disease

Oedema due to hepatic disease

Oedema due to renal disease

Oedema mucosal


#### Oedema neonatal

Oedema peripheral

Oedematous kidney

Oesophageal oedema

Oropharyngeal oedema

Pelvic fluid collection

Pericardial effusion

Perinephric collection

Perinephric oedema

Peripheral oedema neonatal

Peripheral swelling

Pleural effusion

Prevertebral soft tissue swelling of cervical space

Pulmonary congestion

Pulmonary oedema

Pulmonary oedema neonatal

Reexpansion pulmonary oedema

Retroperitoneal effusion

Retroperitoneal oedema

Scleroedema

Skin oedema

Skin swelling

Spinal cord oedema

Subdural effusion

Swelling

Testicular swelling

Vasogenic cerebral oedema

Visceral oedema

#### Excluded PTs

Administration site joint effusion

Administration site oedema

Administration site swelling

Application site joint effusion

Application site joint swelling

Application site oedema

Application site swelling

Catheter site oedema

Implant site oedema

Implant site swelling

Incision site oedema

Incision site swelling

Infusion site joint effusion

Infusion site joint swelling

Infusion site oedema

Infusion site swelling


Statistical Analysis Plan EDMS-RIM-297091

Injection site joint swelling
Injection site oedema
Injection site swelling
Instillation site oedema
Medical device site joint effusion
Medical device site joint swelling
Puncture site oedema
Vaccination site joint effusion
Vaccination site joint swelling

#### 3 ANEMIA/HEMOGLOBIN DECREASE

AEs are included in this grouping if they contain an event Preferred Term (PT) within either of the following Standardised MedDRA Queries (SMQs): 'Haematopoietic erythropenia', or 'Haematopoietic cytopenias affecting more than one type of blood cell' (with the exception of 2 unspecific PTs: 'Blood disorder', 'Blood count abnormal'), or if they contain an event with any MedDRA PT containing the text 'anaemia', i.e., any of the following MedDRA PTs:

Anaemia

Anaemia folate deficiency

Anaemia Heinz body

Anaemia macrocytic

Anaemia megaloblastic

Anaemia neonatal

Anaemia of chronic disease

Anaemia of malignant disease

Anaemia of pregnancy

Anaemia postoperative

Anaemia prophylaxis

Anaemia splenic

Anaemia vitamin B12 deficiency

Anaemia vitamin B6 deficiency

Aplasia pure red cell

Aplastic anaemia

Aspiration bone marrow abnormal

Autoimmune anaemia

Autoimmune aplastic anaemia

Autoimmune haemolytic anaemia

Autosomal recessive megaloblastic anaemia


Statistical Analysis Plan EDMS-RIM-297091

#### Bicytopenia

Biopsy bone marrow abnormal

Blood incompatibility haemolytic anaemia of newborn

Blood loss anaemia

Blood loss anaemia neonatal

Bone marrow disorder

Bone marrow failure

Bone marrow infiltration

Bone marrow myelogram abnormal

Bone marrow necrosis

Bone marrow toxicity

Cardiac haemolytic anaemia

Cold type haemolytic anaemia

Congenital anaemia

Congenital aplastic anaemia

Congenital dyserythropoietic anaemia

Coombs negative haemolytic anaemia

Coombs positive haemolytic anaemia

Cytopenia

Deficiency anaemia

Erythroblast count abnormal

Erythroblast count decreased

Erythroid maturation arrest

Erythropenia

Erythropoiesis abnormal

Febrile bone marrow aplasia

Foetal anaemia

Full blood count decreased

Gelatinous transformation of the bone marrow

Haematocrit abnormal

Haematocrit decreased

Haematotoxicity

Haemoglobin abnormal

Haemoglobin decreased

Haemolytic anaemia

Haemolytic anaemia enzyme specific

Haemolytic icteroanaemia

Hand and foot syndrome secondary to sickle cell anaemia


Hereditary haemolytic anaemia

Hereditary sideroblastic anaemia

Hexokinase deficiency anaemia

Hyperchromic anaemia

Hypochromic anaemia

Hypoplastic anaemia

Immune-mediated pancytopenia

Iron deficiency anaemia

Leukoerythroblastic anaemia

Melanaemia

Microangiopathic haemolytic anaemia

Microcytic anaemia

Myelodysplastic syndrome

Myelodysplastic syndrome transformation

Myelofibrosis

Myeloid metaplasia

Nephrogenic anaemia

Normochromic anaemia

Normochromic normocytic anaemia

Normocytic anaemia

Pancytopenia

Panmyelopathy

Pernicious anaemia

Plasmablast count decreased

Primary myelofibrosis

Proerythroblast count abnormal

Proerythroblast count decreased

Protein deficiency anaemia

Pyruvate kinase deficiency anaemia

Red blood cell count abnormal

Red blood cell count decreased

Refractory anaemia with an excess of blasts

Refractory anaemia with ringed sideroblasts

Reticulocyte count abnormal

Reticulocyte count decreased

Reticulocyte percentage decreased

Reticulocytopenia

Scan bone marrow abnormal


Statistical Analysis Plan EDMS-RIM-297091

Sickle cell anaemia
Sickle cell anaemia with crisis
Sideroblastic anaemia
Spherocytic anaemia
Spur cell anaemia
Warm type haemolytic anaemia

#### 4 HYPOTENSION

AEs are included in this grouping if their coded PTs are included in the following list of PTs:

Blood pressure ambulatory decreased, Blood pressure decreased, Blood pressure diastolic decreased, Blood pressure orthostatic decreased, Blood pressure systolic decreased, Diastolic hypotension, Hypotension, Mean arterial pressure decreased, Orthostatic hypotension, Procedural hypotension.


Statistical Analysis Plan EDMS-RIM-297091

# Appendix D Discussion and further considerations of the applied statistical methods

NA


#### Appendix E Protocol deviation code list

## **Document Revision History:**



## Appendix F. Outputs and SAS code for KM estimates

The LIFETEST SAS procedure in t-t2dth\_sas.txt is used for the computation of the estimates. A selection of the relevant part of code to generate the results for the cohort Macitentan 10mg (DB/OL) is shown below for illustrative purposes with further elucidation for clarity:

```
data d1:
  set adam.addeath;
  where (saf1fl='Y' or saf2fl='Y');
proc sort data=d1 nodupkey;
  by usubjid cestdt;
run;
proc lifetest data=d1
    method=KM
    alphaqt=0.05
    CONFTYPE=loglog
    plots=survival(atrisk=0 to 126 by 6)
    outsurv=sci 1(rename=( censor =censor))
    timelist=0 6 12 18 24 30 36 42 48 54 60 66 72 78 84 90 96 102 108 114 120 126;
    time ttd1*cnsr(1);
    by pool1fl;
    where pool1fl='Y' and saf1fl='Y';
 run;
```

TPL-000241 v02

Macitentan (JNJ-67896062/ACT-064992) AC-055-303

## E


Statistical Analysis Plan EDMS-RIM-297091


The key elements for the analysis are:

i) Dataset ADDEATH included in

## ii) ADDEATH variables:

POOL1FL, SAF1FL for the selection of safety set in the cohort 10mg DB/OL data POOL2FL, SAF2FL for the selection of safety set in the cohort 10mg OL data

TTD1 time to death in months for DB/OL cohort TTD2 time to death in month for OL cohort CNSR that is 0 for events and 1 for censoring

iii) Documentation: a full description of the datasets and variables including source and derivation is included in the define.xml and define.pdf

Macitentan (JNJ-67896062/ACT-064992) AC-055-303 21 December 2020, page 69/69


Statistical Analysis Plan EDMS-RIM-297091

# Document history

| Version | Effective Date | Reason |
|-----------|----------------|--------|
| Final 1.0 | 21-Dec-2020 | |